CLINICAL TRIAL: NCT03841877
Title: Color Dental Alteration Caused by Endodontic Treatment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: There were not participants to complete sample size
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Noéli Boscato, PhD, Professor, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUfpel 2
Record Dates: First submitted 2018-11-11; First posted 2019-02-15 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Endodontically Treated Teeth; Tooth Discoloration; Root Canal Infection
MeSH Terms: conditions — Tooth, Nonvital; Tooth Discoloration | interventions — Endodontics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AH Plus-Cervical (Experimental): The objective is evaluate the color change (ΔE00) originated from epoxy resin (AH Plus) endodontic sealer, sectioned at the cervical level.
  The ΔE00 will be evaluated using the measurements data obtained in a period between the immediate endodontic treatment versus after 3, 6 and 12 months.
  The values of ΔE00 obtained for each sealer, cut and time will be analyzed by multifactorial analysis to verify associations of the outcomes with the ΔE00.
  Interventions: Procedure: endodontic treatment
- MTA Fillapex-Cervical (Experimental): The objective is evaluate the color change (ΔE00) originated from mineral trioxide aggregate (MTA Fillapex) endodontic sealer, sectioned at the cervical level.
  The ΔE00 will be evaluated using the measurements data obtained in a period between the immediate endodontic treatment versus after 3, 6 and 12 months.
  The values of ΔE00 obtained for each sealer, cut and time will be analyzed by multifactorial analysis to verify associations of the outcomes with the ΔE00.
  Interventions: Procedure: endodontic treatment
- AH Plus-2mm (Experimental): The objective is evaluate the color change (ΔE00) originated from epoxy resin (AH Plus) endodontic sealer, sectioned 2 mm below cervical level.
  The ΔE00 will be evaluated using the measurements data obtained in a period between the immediate endodontic treatment versus after 3, 6 and 12 months.
  The values of ΔE00 obtained for each sealer, cut and time will be analyzed by multifactorial analysis to verify associations of the outcomes with the ΔE00.
  Interventions: Procedure: endodontic treatment
- MTA Fillapex-2mm (Experimental): The objective is evaluate the color change (ΔE00) originated from mineral trioxide aggregate (MTA Fillapex) endodontic sealer, sectioned 2 mm below cervical level.
  The ΔE00 will be evaluated using the measurements data obtained in a period between the immediate endodontic treatment versus after 3, 6 and 12 months.
  The values of ΔE00 obtained for each sealer, cut and time will be analyzed by multifactorial analysis to verify associations of the outcomes with the ΔE00.
  Interventions: Procedure: endodontic treatment

INTERVENTIONS:
Procedure: endodontic treatment — The operator will remove the pulp inside the tooth, clean, disinfect and shaping the root canals and seal the space with endodontic sealer.

SUMMARY:
The color change of endodontically treated teeth is a common concern in clinical practice. The objective of this study will be to evaluate, in vivo, the color change (ΔE00) caused by endodontic treatment. A randomized clinical trial (RCT) will be conducted with the objective of evaluating ΔE00 originated from epoxy resin (AH Plus) and mineral trioxide aggregate (MTA Fillapex) endodontic sealers, sectioned at the cervical level and 2 mm below, in a period between the immediate endodontic treatment versus after 3, 6 and 12 months.

DETAILED DESCRIPTION:
The sample syze determined that 48 anterior teeth (incisors and canines) and posterior teeth (premolars) should be included in the study. The sealer and cut will be randomly determined at time of endodontic treatment, originating four groups (n = 12): AH Plus-Cervical, MTA Fillapex-Cervical, AH Plus-2mm and MTA-2mm. The endodontic access cavities will be sealed with resin composed of the color of the dental element. The mean, standard deviation and confidence interval (CI 95%) of the values of ΔE00 obtained for each sealer will be initially analyzed using the variable cut level (cervical or 2mm) using the T test. Indeed, the values of ΔE00 will be analyzed by two-way analysis of variance, where the level of the cut and the type of sealer will be the factors under study.

ELIGIBILITY:
Inclusion Criteria:

endodontically treated tooth, without intraradicular retainer and fixation;

* presence of homologous tooth to that treated, with pulp vitality and at least 1/3 of the crown;
* correctly patient's file showing the endodontic treatment day, the endodontic filler used, the pulp condition at the first consultation, and periapical radiography, obtained with the use of a radiographic positioner, preserved and with a clear apical image

Exclusion Criteria:

* dental elements submitted to retreatment;
* files with insufficient data, and absence of quality periapical radiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Color change | After immediate endodontic treatment versus after 3, 6 and 12 months
  Color alteration will be evaluated using the measurements obtained in the homologous tooth (without endodontic treatment) versus the measurement obtained from the tooth treated endodontically. Data will be analyzed according to sealer, cut and time

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Pelotas, Pelotas, Rio Grande do Sul, Brazil